CLINICAL TRIAL: NCT05575947
Title: A Comparative Analysis of da Vinci-Assisted and Laparoscopic Duodenal Switch (DS) Bariatric Surgical Procedures
Brief Title: Comparative Analysis of da Vinci-Assisted and Laparoscopic Duodenal Switch Bariatric Surgical Procedures
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: Bariatric Surgery
Record Dates: First submitted 2022-09-20; First posted 2022-10-12 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- robotic-assisted: Robotic-assisted cases converted to open will be part of the robotic cohort.
  Comparison of the following safety and effectiveness related surgical outcomes across robotic-assisted and laparoscopic cohorts:
  Safety Related Outcomes
  1. Intraoperative Complication Rates
  2. Transfusion Rates
  3. 30-Day Post-Operative Complication Rates
  4. 30-Day Readmission Rates
  5. 30-Day Reoperation Rates
  6. 30-Day Mortality
  Effectiveness Related Outcomes
  1. Conversion Rate to Open Surgery
  2. Operative Time
  3. Length of Hospital Stay
  Interventions: Device: da Vinci Surgical System
- laparoscopic: Laparoscopic cases converted to open will be part of the laparoscopic cohort.
  Comparison of the following safety and effectiveness related surgical outcomes across robotic-assisted and laparoscopic cohorts:
  Safety Related Outcomes
  1. Intraoperative Complication Rates
  2. Transfusion Rates
  3. 30-Day Post-Operative Complication Rates
  4. 30-Day Readmission Rates
  5. 30-Day Reoperation Rates
  6. 30-Day Mortality
  Effectiveness Related Outcomes
  1. Conversion Rate to Open Surgery
  2. Operative Time
  3. Length of Hospital Stay
  Interventions: Procedure: laparoscopic bariatric surgery

INTERVENTIONS:
Device: da Vinci Surgical System — da Vinci Surgical System
  Groups: robotic-assisted
Procedure: laparoscopic bariatric surgery — laparoscopic bariatric surgery
  Groups: laparoscopic

SUMMARY:
To compare the safety and effectiveness of robotic-assisted Duodenal-Switch Bariatric Surgical Procedures (including Biliopancreatic Diversion-Duodenal-Switch/BPD-DS, Single Anastomosis- Duodeno Ileal Bypass with Sleeve/SADI-S, and One Anastomosis Duodenal Switch/OADS) with laparoscopic approaches using real world data (RWD) from the Premier Healthcare Database (PHD).

DETAILED DESCRIPTION:
To compare the safety and effectiveness of robotic-assisted Duodenal-Switch Bariatric Surgical Procedures (including Biliopancreatic Diversion-Duodenal-Switch/BPD-DS, Single Anastomosis- Duodeno Ileal Bypass with Sleeve/SADI-S, and One Anastomosis Duodenal Switch/OADS) with laparoscopic approaches using real world data (RWD) from the Premier Healthcare Database (PHD). The study endpoints include:

Safety Related Outcomes

1. Intraoperative Complication Rates
2. Transfusion Rates
3. 30-Day Post-Operative Complication Rates*
4. 30-Day Readmission Rates*
5. 30-Day Reoperation Rates*
6. 30-Day Mortality*

Effectiveness Related Outcomes

1. Conversion Rate to Open Surgery
2. Operative Time
3. Length of Hospital Stay

ELIGIBILITY:
Inclusion Criteria-

1. Patients who are ≥ 18 years old and had a primary laparoscopic or robotic-assisted bariatric surgery procedure with a duodenal switch (DS) defined herein as BPD-DS, SADI-S, or OADS; and,
2. Met one of the below qualifications:

   * Body mass index (BMI) > 40 kg/m2 OR
   * BMI > 35 kg/m2 and had one of the following obesity-related co-morbidities such as type II diabetes mellitus, hypertension, sleep apnea and other respiratory disorders, non-alcoholic fatty liver disease, osteoarthritis, lipid abnormalities, gastrointestinal disorders, or heart disease according to the US Centers of Medicare & Medicaid Services (CMS) criteria for the use of bariatric surgery in adults

Exclusion Criteria-

* Were diagnosed with cancer; or
* Underwent an outpatient DS bariatric surgical procedure; or
* Underwent an emergent DS bariatric surgical procedure; or
* Underwent a DS procedure concomitant to a different primary procedure (i.e., colon resection)
* Underwent a revisional DS bariatric surgical procedure (i.e., patient had a prior bariatric procedure within three (3) years of the DS procedure)
* Have missing operating room (OR) time data (i.e., incomplete billing record)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion/exclusion criteria iwho underwent DS Bariatric Surgical Procedures between January 1, 2016 and December 31, 2020 will be included. Acute and 30-day follow up data will be included in this analysis.
Sampling Method: Probability Sample
Enrollment: 1878 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Intraoperative Complication Rates (Safety) | Intraoperative
  Incidence of complications occuring intraoperatively
Transfusions (Safety) | perioperative
  Transfusion Rates Rate of transfusion that occur intraoperatively and postoperatively
30-Day Post-Operative Complication Rates (Safety) | Intraoperative to 30-days (from the date of surgery upto 30-days)
  Incidence of complications that occur after surgery to 30-days
30-Day Readmission Rates (Safety) | Upto 30 days
  Incidence of readmission that occur after discharge
30-Day Reoperation Rates (Safety) | upto 30 days following the documented date of the surgery
  Incidence of reoperations that occur after till 30 days
30-day Mortality Rate (Safety) | Intra-operative to 30-days
  Incidence of mortality until 30 days
Conversion rate to open surgery (Effectiveness) | Intraoperative
  Incidence of conversion to open that occur intraoperatively
Operative Time (Effectiveness) | Intraoperative
  Amount of time it takes to complete the procedure (in min)
Length of hospital Stay (Effectiveness) | perioperative
  Number of days participant is in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Usha L Kreaden, Study Director — Intuitive Surgical
Locations (1):
- Intuitive Surgical, Sunnyvale, California, United States